CLINICAL TRIAL: NCT03846206
Title: Changes in Bacterial Translocation and Immune Activation in Patients Infected With HIV After Change to a Supplemented Mediterranean Diet: Two Arms Randomized Prospective Trial.
Brief Title: Mediterranean Diet and Bacterial Translocation and Immune-activation in Patients With HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Felipe Garcia, DOCTOR, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clinic Hospital of Barcelona
Record Dates: First submitted 2017-06-14; First posted 2019-02-19 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Hiv
Keywords: Microbiota.; Mediterranean Diet; Bacterial Traslocation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: . One hundred and two patients who will be randomized to continues usual diet or to a Mediterranean diet supplemented with 50 g / day of olive oil and 15g / day of nuts for three months. Throughout the study a specialized dietician will monitor the patients. Blood samples will be collected to assess parameters of bacterial translocation, inflammation and immune activation. To assess compliances with diet, urine samples will be collected too, and stool samples to study changes in gut microbiota. All the samples will be collected at the beginning and 90 days after the inclusion in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mediterranean diet (Experimental): Patients do Mediterranean diet supplemented with 50 g / day of olive oil and 15g / day of nuts for three months
  Interventions: Dietary Supplement: mediterranean diet
- Usual diet (No Intervention): Patients do usual diet for three months

INTERVENTIONS:
Dietary Supplement: mediterranean diet — a Mediterranean diet supplemented with 50 g / day of olive oil and 15g / day of nuts for three months
  Arms: mediterranean diet

SUMMARY:
Evaluate if a change to a Mediterranean diet supplemented with nuts and olive oil decreases bacterial translocation and immune activation by a change in the microbiome in successfully treated HIV-1 infected patients with CD4> 500cells/ml.

DETAILED DESCRIPTION:
Mediterranean diet supplemented by nuts and extra virgin olive oil has shown to reduce mortality, cardiovascular diseases, and breast cancer in HIV uninfected individuals. It is likely that changes in the microbiome could play a role in this effect. The goal of the study is to evaluate if a change to a Mediterranean diet supplemented with nuts and olive oil decreases bacterial translocation and immune activation by a change in the microbiome in successfully treated HIV-1 infected patients with CD4> 500cells/ml. One hundred and two patients who will be randomized to continues usual diet or to a Mediterranean diet supplemented with 50 g / day of olive oil and 15g / day of nuts for three months. Throughout the study a specialized dietician will monitor the patients. Blood samples will be collected to assess parameters of bacterial translocation, inflammation and immune activation. To assess compliances with diet, urine samples will be collected too, and stool samples to study changes in gut microbiota. All the samples will be collected at the beginning and 90 days after the inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age;
* To sign voluntary informed consent;
* Male or female patients with a negative pregnancy test before inclusion in the study;
* Proven HIV infection (with HIV-1 positive antibodies);
* Patient should be on stable treatment with cART for at least 1 year
* The mean of all CD4 measurements during the year prior to the initiation of cART should be equal to greater than 350 cells / mm3
* The number of CD4 + at the time of recruitment must be equal to or greater than 500 cells / mm3;
* HIV viral load should be undetectable at least 6 months prior to study inclusion, and less determinations (occasional blips above the undetectable level are allowed).

Exclusion Criteria:

* Acquired Immunodeficiency Syndrome.
* Active opportunistic diseases.
* Patients coinfected with HCV or HBV
* Coagulopathy
* Renal insufficiency (creatinine> 1.5 mg / dL)
* Pregnancy or breastfeeding
* Inability to sign informed consent
* Active opportunistic infections, or any active infection or cancer within 30 days prior to the screening visit;
* Therapy with immunomodulatory agents, including cytokines (eg IL-2) and gammaglobulins or chemotherapy within 90 days prior to the screening visit;
* Use of anticoagulant medication;
* Use of any type of experimental medication during the 90 days prior to study entry;
* Uncontrolled psychiatric disorder;
* Patients with uncontrolled active autoimmune diseases;
* Usual use of antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2016-07-01; Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Differences in levels of sCD14 at baseline and month 3 between groups | 2 year
  parameters of bacterial translocation

SECONDARY OUTCOMES:
Changes in EndocAB and LBP levels at baseline and month 3 between groups. | 2 year
  other parameters of bacterial translocation.
Changes in microbiota (fecal 16s rRNA) at baseline and month 3 between groups | 2 years
  Microbioma
Changes in ultrasensitive PCR, TNF-alpha, IL-6 and Dimer-D at baseline and month 3 between groups | 2 years
  inflammatory markers
Changes in lipids at baseline and month 3 between groups | 2 years
  Lipids
Changes in expression of CD38, HLA DR in CD4 and CD8 T cells at baseline and month 3 between groups | 2 years
  immune-activation markers
Changes in total and integrated DNA | 2 years
  Marker of HIV reservoir

CONTACTS AND LOCATIONS:
Overall Officials: Felipe García, MD, PhD, Principal Investigator — Institut d'Investigacions Biomèdiques August Pi i Sunyer
Locations (1):
- Felipen Garcia, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No